CLINICAL TRIAL: NCT04512625
Title: Efficacy of Three Commercially Available Desensitizers in Reducing Post Tooth Preparation Sensitivity for a Fixed Dental Prosthesis- A Randomized Controlled Clinical Trial.
Brief Title: Desensitizers in Reducing Post Tooth Preparation Sensitivity for a Fixed Dental Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Dr Harisha Dewan, Assistant Professor, University of Jazan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UJazan
Record Dates: First submitted 2020-08-10; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Dentin Hypersensitivity
Keywords: Pre-cementation sensitivity, Desensitizers
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: The present study was designed as a single-center, parallel, double-blind, randomized, controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The application of the stimuli and the desensitizers and collection of subjects' responses during the visits was carried out by two well-trained examiners. After providing informed consent, the first examiner allocated a number to each patient. The patients were blinded to whether they were in the control group or one of the desensitizer groups. The application of the agents was also carried out by the same examiner. The tests were carried out by the second examiner who also recorded the sensitivity during the visits. Group allotment and the application of the agents were thus carried out by the first examiner, which were concealed from the second examiner who assessed and recorded the sensitivity scores, making the study double-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Control group (No Intervention): Sensitivity level scores were evaluated on the Visual Analogue Scale using cold stimuli (Cold Test) and electrical stimuli (Electric Pulp Test) at all the 3-time intervals, i. e first, second, and the third visit and then telephonically two weeks after the final cementation.
- Group GL (Gluma desensitizer) (Experimental): In desensitizer groups, respective desensitizer application was done following the manufacturer's directions immediately after tooth preparation before final impressions were made (first visit), before metal try-in (second visit) and before final cementation (third visit). Sensitivity level scores were evaluated, before the desensitizer application, on the Visual Analogue Scale using cold stimuli (Cold Test) and electrical stimuli (Electric Pulp Test) at all the 3-time intervals, i. e first, second, and the third visit and then telephonically two weeks after the final cementation. The data were statistically analyzed using one-way ANOVA followed by post-hoc Bonferroni and unpaired t-test.
  Interventions: Biological: Desensitizers
- Group SF (SheildForce desensitizer) (Experimental): In desensitizer groups, respective desensitizer application was done following the manufacturer's directions immediately after tooth preparation before final impressions were made (first visit), before metal try-in (second visit) and before final cementation (third visit). Sensitivity level scores were evaluated, before the desensitizer application, on the Visual Analogue Scale using cold stimuli (Cold Test) and electrical stimuli (Electric Pulp Test) at all the 3-time intervals, i. e first, second, and the third visit and then telephonically two weeks after the final cementation. The data were statistically analyzed using one-way ANOVA followed by post-hoc Bonferroni and unpaired t-test.
  Interventions: Biological: Desensitizers
- Group TS (Telio CS desensitizer) (Experimental): In desensitizer groups, respective desensitizer application was done following the manufacturer's directions immediately after tooth preparation before final impressions were made (first visit), before metal try-in (second visit) and before final cementation (third visit). Sensitivity level scores were evaluated, before the desensitizer application, on the Visual Analogue Scale using cold stimuli (Cold Test) and electrical stimuli (Electric Pulp Test) at all the 3-time intervals, i. e first, second, and the third visit and then telephonically two weeks after the final cementation. The data were statistically analyzed using one-way ANOVA followed by post-hoc Bonferroni and unpaired t-test.
  Interventions: Biological: Desensitizers

INTERVENTIONS:
Biological: Desensitizers — The main aims and objectives of the present study were to evaluate and compare the effectiveness of three commercially available desensitizing agents: Gluma (Hareus Kulzer), Sheildforce Plus (Tokuyama), and Telio CS (Ivoclar Vivadent) desensitizer in reducing the pre- and post-cementation sensitivity for full coverage restorations.
  Arms: Group GL (Gluma desensitizer); Group SF (SheildForce desensitizer); Group TS (Telio CS desensitizer)

SUMMARY:
The main purpose of the present study was to evaluate and compare the effectiveness of three kinds of commercially available desensitizing agents: Gluma, Sheildforce plus, and Telio CS desensitizers in reducing the pre- and post-cementation sensitivity for full coverage restorations.

DETAILED DESCRIPTION:
During the first visit, standard prosthodontic principles were followed to prepare the teeth for complete coverage restorations using high-speed handpiece and copious water-coolant spray. After the effect of local anesthesia was worn off, baseline sensitivity (first reading) was recorded on the VAS using Cold Test and Electric Pulp Test (EPT) . Final impression using addition silicon (Virtual from Ivoclar Vivadent, Amherst, NY) was made, and the provisional prosthesis was fabricated using Protemp TM II (3M ESPE, Germany), by the direct method using polyvinyl siloxane putty (ExpressTM STD, 3M ESPE) matrix. The first application of desensitizer was done then on the desensitizer group according to the manufacturer's recommendation. The fabricated provisional prosthesis was cemented with non-eugenol provisional cement Tempbond NE (Rely XTM TempNE, 3M ESPE, Germany) and the patient was recalled for the metal try-in. During the second visit, the provisional prosthesis was removed and the patient's response to Cold Test and EPT was again recorded on VAS (second reading) and the metal try-in was carried out. The second application of desensitizing agent was done, the provisional prosthesis was re-cemented, and the patient was recalled for final cementation. During the third visit, the provisional prosthesis was removed, the patient's response to Cold Test and EPT was again recorded (third reading), and the third application of desensitizing agent was done before cementing the final prosthesis with G-cem resin cement. The control group had similar clinical steps except for the application of desensitizer, Evaluation of sensitivity level Subjective evaluation of pain produced by cold and electrical stimulus was done, for checking pre-cementation sensitivity. Before starting the procedure, patients were explained about the Cold Test, EPT, and the VAS scores.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were: minimum of one posterior tooth missing and patient in need of fixed dental prosthesis (porcelain fused to metal); abutment teeth with a vital pulp, normal apical periodontal ligament space, no history of hypersensitivity; and previous restorations not involving more than 50% of the coronal tooth surface.

Exclusion Criteria:

* The exclusion criteria were: patients with chronic diseases, gross oral pathology, or those undergoing any kind of medications; subjects with teeth that had extensive restorations, mobility or periodontal diseases; pregnant or lactating women; and individuals participating in any other clinical study.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Pre-cementation sensitivity | First Visit, 3 hours after preparation.
  Pre-cementation sensitivity is evaluated after Cold Test and EPT using the Visual Analog Scale(1-10, 0 = 'no pain' (non-sensitive) and 10 ='severe pain' (extremely hypersensitive).
Pre-cementation sensitivity | Second Visit, 1 week after tooth preparation.
  Pre-cementation sensitivity level is evaluated after Cold Test and EPT using the Visual Analog Scale(1-10, 0 = 'no pain' (non-sensitive) and 10 ='severe pain' (extremely hypersensitive).
Pre-cementation sensitivity | Third Visit, 1 week after metal try in.
  Pre-cementation sensitivity is evaluated after Cold Test and EPT using the Visual Analog Scale(1-10, 0 = 'no pain' (non-sensitive) and 10 ='severe pain' (extremely hypersensitive).
Post-cementation sensitivity | 2 weeks post cementation.
  Patient's response to sensitivity are evaluated over a telephonic interview.

CONTACTS AND LOCATIONS:
Overall Officials: Harisha Dewan, MDS, Principal Investigator — University of Jazan
Locations (1):
- Harisha Dewan, Jizan, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Currently, there is no plan to share IPD. However, the interested researchers can request it directly to us if the need arises.